CLINICAL TRIAL: NCT01558908
Title: Allogeneic,Unrelated, Menstrual Derived, Mesenchymal Stem Cell-Like, Endometrial Cells; Administered Intramuscular
Brief Title: Phase I/II Trial of Endometrial Regenerative Cells (ERC) in Patients With Critical Limb Ischemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medistem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDS-027
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Peripheral Vascular Diseases
Keywords: critical limb ischemia
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

ARMS (1):
- Intramuscular injection of ERC (Experimental)
  Interventions: Biological: Administration of ERC

INTERVENTIONS:
Biological: Administration of ERC — Patients will be treated with either 25 million, 50 million, or 100 million ERC by intramuscular injection.

SUMMARY:
This is a 15 patient clinical trial assessing the safety and feasibility of using Endometrial Regenerative Cells (ERC) in patients with critical limb ischemia (CLI) that are not eligible for surgical or catheter-based interventions. Three doses of ERC will be examined. The hypothesis is that ERC administration will be well-tolerated and possibly induce a therapeutic benefit.

DETAILED DESCRIPTION:
The purpose of the trial is to determine safety of intramuscularly derived menstrual mesenchymal stem cells (otherwise known as Endometrial Regenerative Cells, or ERC) in patients with critical limb ischemia ineligible for revascularization. Safety will be defined as freedom from treatment associated adverse events. Efficacy parameters will comprise endpoints of changes in ankle-brachial index, toe-brachial index, TcPO2, ulcer healing, rest pain, quality of life, and reduction in amputation.

Patients will receive 25, 50, or 100 million menstrual derived mesenchymal stem cells (Endometrial Regenerative Cells: ERC) in ten injections of 2.5, 5, or 10 million mesenchymal stem cells suspended in a volume of 1 ml per injection. Injections will be spaced at least 2 centimeters apart from each other in the gastrocnemius muscle above the failed vascular perfusion area.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant patients with critical limb ischemia, Rutherford IV-V, manifested as rest pain or tissue loss, or with disabling claudication, manifested as exercise induced thigh or calf pain that impairs activities of daily living, who are not candidates for surgical bypass or angioplasty due to unfavorable arterial anatomy or absence of adequate autogenous vein for a below-knee bypass.
2. Patients over 18 years of age with an expected survival of more than one year after treatment.
3. Unreconstructable arterial disease will be determined by a vascular surgeon who is not participating in the study. Unreconstructable arterial disease is defined by atherocclusive lesions within the arterial tree of the extremity that due to extent or morphology are not amenable to surgical bypass or PTCA and stenting.
4. Patients with a maximum of 3 non-healing 'flat' surface or 'transdermal' ulcers Grades 1-2, no ulcer bigger than 2 centimeters (2)
5. Patients with unfavorable anatomy or who are medically unfit to undergo bypass as determined by a vascular surgeon who is not participating in the study.
6. Vascular imaging (eg angiogram or MRA) to determine vascular anatomy must be conducted within 3 months of study entry.
7. Patients with low/absent perfusion in the area at or below the gastrocnemius muscle
8. Objective evidence of severe peripheral arterial disease will include an ankle brachial index (ABI) of less than 0.55, and/or a resting toe brachial index (TBI) of less than 40.
9. Patients must be competent to give consent.
10. No history of malignant disease except for nonmelanoma skin cancer, no suspicious findings on chest x-ray, mammography (women over age 35) , Papanicolaou smear (women over age 40), a normal fecal occult blood (over age 50) and a normal prostate specific antigen (men over age 45).
11. Patients must have a prothrombin Time (PT) between 12-14 seconds, a partial thromboplastin time (PTT) of 18-28 seconds, and platelet count >100,000/microliter
12. Patients must have white blood cell count (4.1-10.9x10(3) cells/µL)
13. Normal liver function tests (AST 8 - 20 U/L, ALT 8 - 20 U/L, and total bilirubin 0.1 - 1.0 mg/dL)
14. Patients must be male or post menopausal women.

Exclusion Criteria:

1. Patients with evidence of active proliferative retinopathy.
2. Patients with poorly controlled diabetes mellitus (HbA1C > 8.5%).
3. Patients with renal insufficiency (Creatinine > 2.5) or failure.
4. Infection as evidenced by WBC count of >15,000 k/cumm and/or temperature >38C.
5. Cellulitis in the afflicted limb that in the opinion of the investigators would require the use of antibiotics or evidence of osteomyelitis corroborated by radiographic or scintigraphic examination.
6. Pregnant women (women capable of childbearing must have a negative pregnancy test)
7. Cognitively impaired adult
8. Lower extremity venous disease with pitting edema.
9. History of organ transplant.
10. Patients with ulcer exudates, dry gangrene or exposed bone.
11. Allergies to beta-lactam antibiotics, amphotericin B, or streptomycin
12. Cardiovascular conditions:

    * Exercise limiting angina (Canadian Cardiovascular Society Class > 3
    * Congestive heart failure (New York Heart Association class > 3
    * Unstable angina
    * Acute ST elevation myocardial infarction (MI) within 1month
    * Transient ischemic attack or stroke within 1 month
    * Severe valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Safety | 52 weeks
  Adverse and serious events recorded

SECONDARY OUTCOMES:
Efficacy | 12 weeks
  Improvements post-treatment in rest pain (VAS), toe pressure and ABI, transcutaneous oximetry and ulcer status (with picture).

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Murphy, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- See also: Murphy et al. Allogeneic endometrial regenerative cells: An "Off the shelf solution" for critical limb ischemia? J Transl Med. 2008 Aug 19;6:45. — http://www.translational-medicine.com/content/pdf/1479-5876-6-45.pdf